CLINICAL TRIAL: NCT03058757
Title: The Effectiveness and Safety of Neoadjuvant Intravesical Mitomycin-C Instillation in Non-muscle Invasive Bladder Cancer Patients: Prospective, Randomized, Phase II Study
Brief Title: The Effectiveness and Safety of Neoadjuvant Intravesical Mitomycin-C Instillation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Ho Kyung Seo, Primary Investigator, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NeoadjMitomycin-C
Record Dates: First submitted 2017-02-15; First posted 2017-02-23 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): No intervention applied.
- Intervention arm (Experimental): neoadjuvant intravesical mitomycin-C 40mg/20ml instillation
  Interventions: Drug: intravesical mitomycin-C 40mg/20ml instillation

INTERVENTIONS:
Drug: intravesical mitomycin-C 40mg/20ml instillation — neoadjuvant Intravesical mitomycin-C 40mg/20ml instillation
  * one day before surgery
  * four hours before surgery
  Other Names: Mitomycin_C Kyowa
  Arms: Intervention arm

SUMMARY:
The aim of this study is to evaluate the effectiveness and safety of neoadjuvant intravesical mitomycin-C instillation in non-muscle invasive bladder cancer patients

DETAILED DESCRIPTION:
Study Design: Intervention Model: Single Group Assignment Masking: Open Label

Primary Outcome Measures:

Recurrence-free survival in neoadjuvant intravesical mitomycin-C 40mg/20ml instillation group and control group.

Secondary Outcome Measures:

Progression-free survival in neoadjuvant intravesical mitomycin-C 40mg/20ml instillation group and control group.

Time to recurrence in neoadjuvant intravesical mitomycin-C 40mg/20ml instillation group and control group.

Change of tumor size after neoadjuvant intravesical mitomycin-C 40mg/20ml instillation.

Safety of neoadjuvant intravesical mitomycin-C 40mg/20ml instillation.

ELIGIBILITY:
Inclusion Criteria:

* The subjects who will undergo transurethral resection of the tumor after diagnosis of bladder cancer
* Male or female aged 18 or over 18 years and not more than 85 years who were diagnosed as bladder cancer
* Normal bone marrow function: Hemoglobin >10 g/dL, ANC >1,500/mm3, platelet count>100,000/mm3
* Normal renal function: serum creatinine ≤ 1.4 mg/dL
* Normal liver function:
* Bilirubin ≤ 1.5 times of upper normal limit
* AST/ALT ≤ 1.8 times of upper normal limit
* Alkaline phosphatase ≤ 1.8 times of upper normal limit
* Subjects who voluntarily decided to participate and signed the written informed consent

Exclusion Criteria:

* Non-urothelial carcinoma
* Muscle invasive bladder cancer
* Subjects who underwent intravesical mitomycin-C instillation after diagnosis of bladder cancer within 3 years
* Prior hypersensitivity reaction history to mitomycin-C
* Neurogenic bladder
* Subjects who underwent chemotherapy due to any cancer within 6 months

Ages: 20 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Recurrence-free survival in neoadjuvant intravesical mitomycin-C 40mg/20ml instillation group and control group. Recurrence will be assessed by CT scan and cystoscopic exam. | 1 year
  Pathologic recurrence free survival after transurethral resection

SECONDARY OUTCOMES:
Progression-free survival in neoadjuvant intravesical mitomycin-C 40mg/20ml instillation group and control group. Progression will be assessed by CT scan. | 1 years
  Pathologic or radiologi progression free survival after transurethral resection
Time to recurrence in neoadjuvant intravesical mitomycin-C 40mg/20ml instillation group and control group. Recurrence will be assessed by CT scan and cystoscopic exam. | 1 years
  Period of from transurethral resection to first pathologic recurrence
Change of tumor size after neoadjuvant intravesical mitomycin-C 40mg/20ml instillation. Change of tumor size will be assessed by CT scan and cystoscopic exam. | 1 years
  Change of tumor size at the time point of diagnostic cystoscope to transurethral resection
Safety of neoadjuvant intravesical mitomycin-C 40mg/20ml instillation. | six years
  Safety will be assessed by International Prostate Symptom Score (IPSS; 0-7, mildly symptomatic; 8-19, moderately symptomatic; 20-35 severely symptomatic) and treatment delay

CONTACTS AND LOCATIONS:
Overall Officials: Ho Kyung Seo, M.D., Principal Investigator — National Cancer Center
Locations (1):
- National Cancer Center, Goyang, South Korea

IPD SHARING:
Plan to Share IPD: No